CLINICAL TRIAL: NCT02006238
Title: A Comparison of Farabloc Fabric With Placebo on Alleviation Hot Flash in Menopausal Women
Acronym: Flash
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H13-03052
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Menopause
Keywords: Hot flash; Farabloc; menopausal women
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Farabloc (Experimental): The participants will sleep on Farabloc fabric nightly for a week.
  Interventions: Device: Farabloc; Device: Nylon Fabric
- Nylon Fabric (Placebo Comparator): The participants will sleep on Nylon fabric nightly for week.
  Interventions: Device: Farabloc; Device: Nylon Fabric

INTERVENTIONS:
Device: Farabloc — The participants will be randomly received Farabloc (experimental) for one week, followed by a 7 day washout and then crossed over to received the Nylon fabric (placebo) for one week.
Device: Nylon Fabric — The participants will be randomly received Nylon fabric (placebo) for one week, followed by a 7 day washout and then crossed over to receive Farabloc (experimental) for one week.

SUMMARY:
This is a prospective, randomized, double-blind, crossover study. The purpose of this study is to determine whether Farabloc fabric is effective in alleviation of hot flash symptoms in menopausal women. This study will require all prospective participants to fill out a week of Hot Flash Diary to determine eligibility before beginning the study. All prospective participants will be assessed for hot flash frequency, hot flash distress and hot flash severity according to their perception in the Hot Flash Diary during the experimental period.

DETAILED DESCRIPTION:
Fifty menopausal volunteers will be randomly assigned to two groups, one receiving Farabloc fabric containing Farabloc (experimental), and the other a similar-appearing fabric made of Nylon (placebo).

All eligible participants will be selected by the initial interview. The following information will be collected during interview process.

* Address
* Medical history
* Concomitant medication
* Allergies

Participants will be asked the following:

1. On a scale from 1 to 10, how much are you bothered by your hot flashes?
2. Do these hot flashes wake you up at night? Around how many times do they occur at night?
3. What are you expectations about this study?

A Menopause Rating Scale questionnaire will be completed by the potential participant to assess symptoms Eligible patients from each group will initially undergo a 7 day washout period before intervention in order to eliminate any effects of hormone replacement therapies (HRT) or herbal supplements that subjects may be using prior to participation in the study. Subjects will be randomized to receive a Farabloc fabric or placebo fabric for one week. After this, the two groups will undergo a second 7 day washout period before crossing over to the other fabric. Once crossed over, participants will use the allocated fabrics for another week.

Participants will be asked not to take their usual HRT or herbal supplements for the entire experimental duration in this study in order to produce impartial, precise and reliable results.

The manufacturer will assign codes for placebo fabric or experimental Farabloc. The randomization code will be broken at the completion of the study for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women with 12 months amenorrhea
* Experiencing more than 2 nocturnal hot flashes nightly.

Exclusion Criteria:

* Other medical conditions associated with night sweats
* Currently on medication associated with night sweats
* Less than 2 nocturnal hot flashes per night
* Allergies to metals
* Abnormal mental status
* MRS scale rating of mild or above
* Currently on hormone replacement therapy or herbal supplements and cannot safety discontinue these for the duration of the study.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of hot flashes | in the past 24 hours
  The number of hot flashes subjects experienced in the past 24 hours

SECONDARY OUTCOMES:
Severity of hot flash | In the past 24 hours
  An overall severity rating of hot flashes using a 10 point numeric scale 0 (not at all ) to 10 (extremely)

CONTACTS AND LOCATIONS:
Overall Officials: York N Hsiang, MB FRCSC, Principal Investigator — University of British Columbia, Division of Vascular Surgery and Vancouver General Hospital
Locations (1):
- Dr. Hsiang's office, 510-943 W. Broadway, Vancouver, British Columbia, Canada